CLINICAL TRIAL: NCT05865301
Title: Outcomes in Pediatric and Young Adult B-Cell Malignancies After Commercially Available Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Pediatric Oncology Experimental Therapeutic Investigators Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-70021; Gift Funding (Other: Bass Center Leukemia Pilot Grant); NCI-2024-06344 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lymphoid Leukemia
Keywords: PRWCC; Foresight
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A (Retrospective data): Participants who have undergone standard of care tisagenlecleucel therapy, Participants will received a questionnaire study using patient reported outcomes.
  Interventions: Other: Questionnaire for patients receiving therapy
- Arm B (Prospective data): Patients enrolled in ARM B will be asked to participate in the biological sample collection. Participants will received a questionnaire
  Interventions: Other: Questionnaire for patients receiving therapy

INTERVENTIONS:
Other: Questionnaire for patients receiving therapy — Questionnaires will be given (at baseline, 1, 3, 6, and 12 months post CAR infusion) including baseline demographics, individual/family and neighborhood socioeconomic data, measures of household material hardship (housing and transportation insecurity, household energy and food insecurity), barriers to care at the CAR T cell institution, as well as patient reported outcomes following Kymriah infusion.

SUMMARY:
To use a consistent and standardized platform to retrospectively and prospectively study children and young adults with B cell malignancies receiving Immunotherapy, blinatumomab and/or inotuzumab ozogamicin.

ELIGIBILITY:
Inclusion Criteria (Arm A)

* Disease Status - B cell precursor acute lymphoblastic leukemia (ALL) or B cell lymphoma

Who either:

* Experienced refractory or relapsed disease, treated with standard chemotherapy, without immunotherapy treatment.

OR

* Previously undergone standard of care immunotherapy with FDA approved therapies, such as Kymriah™ (CTL019, tisagenlecleucel), blinatumomab or

  * Age: Greater than or equal to 0 year of age and less than or equal to 26 years of age.

Inclusion Criteria (Arm B)

* Disease Status - B cell precursor acute lymphoblastic leukemia (ALL) or B cell lymphoma
* Age: Greater than or equal to 0 year of age and less than or equal to 26 years of age
* Patients who are either:

  * Undergoing evaluation for leukapheresis for planned standard of care tisagenlecleucel therapy, or planned for therapy with blinatumomab or inotuzumab. (Patients who received prior tisagenlecleucel, blinatumomab or inotuzumab on an established clinical trial and are now scheduled for commercial CAR, blinatumomab or inotuzumab therapy are also eligible) Or
  * Experienced refractory or relapsed B cell precursor acute lymphoblastic leukemia (ALL) or B cell lymphoma
* Ability to give informed consent. All subjects ≥ 18 years of age must be able to give informed consent or have legal authorized representative (LAR) (i.e. parent or guardian) to consent, if not in capacity to give consent independently. For subjects <18 years old their LAR must give informed consent. Pediatric subjects will be included in age appropriate discussion and written assent will be obtained for those > 7 years of age, when appropriate, according to institutional procedures.

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Both Arm A and Arm B, includes retrospective and prospective data collection for patients experiencing refractory disease or first relapse, who have not received immunotherapy and are not yet being considered for immunotherapy. Retrospective data collection will parallel Arm A and patients will not require consent or assent. Prospective data collection will parallel Arm B and will require patient consent and assent as relevant
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
WECARE-Survey | at baseline
  Participant will take part in a one-time questionnaire to address CAR specific questions.
  WECARE survey, consists of questions used to identify seven unmet material needs (education, employment, food security, housing, childcare, household heat, language)
Retrospective WECARE Survey | up to 12 months post infusion
  Surveys will be administered at a single time point post-CAR

SECONDARY OUTCOMES:
overall survival (OS) | at baseline up to 12 months post infusion
  Overall survival was the duration from the start of study treatment to death.
event-free-survival (EFS) | at baseline up to 12 months post infusion
  probability of recurrence or progression of in patients
duration of remission (DOR) | at baseline up to 12 months post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Liora Schultz, M.D, Principal Investigator — Stanford University
Locations (21):
- United States (21):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford University, Palo Alto, California
  - UCSF (Benioff Children's), San Francisco, California
  - Nemours Children's Hospital, New Castle, Delaware
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Louis Children's (Washington University), St Louis, Missouri
  - Children's Hospital at Montefiore, The Bronx, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Saint Jude Children's Research Hospital, Fairfax, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin